CLINICAL TRIAL: NCT03963362
Title: Clinical Study to Evaluate Pharmacokinetics of GLA5PR Tablet According to the Renal Function
Brief Title: The Pharmacokinetics of GLA5PR Tablet According to the Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLA5PR-107
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Neuropathic Pain
Keywords: GLA5PR; Renal function; Pharmacokinetics; Pregabalin
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Administration of GLA5PR 75 mg as 60~89 mL/min (Experimental): Administration of GLA5PR 75 mg as 60~89 mL/min(CLcr)
  Interventions: Drug: GLA5PR tablet 75 mg
- Administration of GLA5PR 75 mg over 90 mL/min (Experimental): Administration of GLA5PR 75 mg over 90 mL/min(CLcr)
  Interventions: Drug: GLA5PR tablet 75 mg
- Administration of GLA5PR 150 mg as 60~89 mL/min (Experimental): Administration of GLA5PR 150 mg as 60~89 mL/min(CLcr)
  Interventions: Drug: GLA5PR tablet 150 mg
- Administration of GLA5PR 150 mg over 90 mL/min (Experimental): Administration of GLA5PR 150 mg over 90 mL/min(CLcr)
  Interventions: Drug: GLA5PR tablet 150 mg
- Administration of GLA5PR 75 mg as 30~59 mL/min (Experimental): Administration of GLA5PR 75 mg as 30~59 mL/min(CLcr)
  Interventions: Drug: GLA5PR tablet 75 mg

INTERVENTIONS:
Drug: GLA5PR tablet 75 mg — GLARS-NF3 tablet
  Arms: Administration of GLA5PR 75 mg as 30~59 mL/min; Administration of GLA5PR 75 mg as 60~89 mL/min; Administration of GLA5PR 75 mg over 90 mL/min
Drug: GLA5PR tablet 150 mg — GLARS-NF3 tablet
  Arms: Administration of GLA5PR 150 mg as 60~89 mL/min; Administration of GLA5PR 150 mg over 90 mL/min

SUMMARY:
To evauate pharmacokinetics of GLA5PR tablet according to the renal function

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject who, at the time of screening, are the age between 19 and 64 years
* Subject who has body weight more than 50 kg (45 kg in women), and less than 80 kg
* Subject who normal renal function of the creatinine clearance calculated by Cockcroft-Gault equation over 90 mL/min
* Subject who the mild renal function of the creatinine clearance between 60 and 89 mL/min calculated by Cockcroft-Gault equation
* Subject who the moderate renal patient of the creatinine clearance between 30 and 59 mL/min calculated by Cockcroft-Gault equation
* Subject who is clinically no significant by a medical history, physical, and psychological examination
* Subject who clinically no significant a vital sign with Investigator's judgment
* Subject who has result of diagnostic laboratory test excluding the items described in exclusion criteria of the 13, and 14, and judged to be clinically no significant when medically by investigator
* Subject who has consented to use a combination of effective contraceptive methods or medically appropriate contraceptive methods from the first administration of the clinical trial drug to the end of the clinical trial (when testing for final safety evaluation) and not to provide sperm or egg
* Subject who is negative the serum and urine hCG test, and is not to pregnant and feeding
* Subject who signed and dated the informed consent form after understanding fully to hear a detailed explanation in the clinical trial
* Subject who is accept to the post-study visit and to be willing to providing of collection the blood, and urine

Exclusion Criteria:

* Subject who is any history of gastrointestinal disease (e.g., Crohn's disease, and others), and surgery (except for simple appendectomy or repair of a hernia), which can influence the absorption of investigational products
* Subject who has a history of hypersensitivity or clinically significant hypersensitivity reactions to drugs or other drugs (aspirin, antibiotics, etc.) that contain components of the clinical trial drug or components of the same class (except for inactive allergic rhinitis)
* Subject who is genetic problem such as galactose intolerance, or Lapp lactose dehydrogenase deficiency, or glucose-galactose uptake disorder
* Subject with the exclusion criteria of 1 to 3, or a significant disease (epilepsy, etc.) and past disease that is considered difficult to participate in clinical trials according to the investigator's judgement
* Subject who had whole blood donation within 60 days or component blood donation within 30 days before the first administration of the investigational product, or transfusion within 60 days before the first administration
* Subject who has participated in any other clinical trials and had medication within 180 days prior to the first administration of investigational product
* Subject who has taken any ethical-the-counter drug or has taken any over-the-counter drug within 14 days before the screening visit, except to the taken the prior-medication for the disease treatment
* Subject who has taken any oriental medicines or any dietary supplements within 30 days, before the screening visit
* Subject who has taken any heavy drinking within 30 days before the screening visit (>21 units/week)
* Subject who has taken a food expected to have an effect on the clinical trial within 7 days, before the screening visit; The food of contained in caffeine (> 2 times/day) The products containing grapefruit (> 2 times/day)
* Subject who has shown positive reaction to drugs that may be abused from a urine drug screening
* Subject who is positive result in smoking or urine nicotine test within 30 days, before the screening visit
* Subject who is positive result in serum test (hepatitis type B test, hepatitis type C test, Human Immunodeficiency Virus (HIV) test, and syphilis test), during the screening period
* Subject who showed the following findings in the tests conducted during the screening period;
* Less than the lower normal limit (LNL) in the Hb.
* In excess of 1.5 times the upper normal limit (UNL) in the hepatic enzyme (AST and ALT), and the alkaline phosphatase values
* In excess of 1.5 times the upper normal limit (UNL) in the total bilirubin
* Subject who is QTc > 450 msec in ECG or a clinically significant abnormal rhythm during the screening period
* Subject who is not eligible person for the clinical trial according to the investigator's judgment

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
The Cmax of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, and 72 hours after administration
  Cmax
The AUClast of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, and 72 hours after administration
  AUClast

SECONDARY OUTCOMES:
tmax of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72 hours after administration
  tmax
t1/2beta of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, and 72 hours after administration
  t1/2beta
AUCinf of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, and 72 hours after administration
  AUCinf
CL/F of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, and 72 hours after administration
  CL/F
Vz/F of Pregabalin | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, and 72 hours after administration
  Vz/F

CONTACTS AND LOCATIONS:
Overall Officials: Minchang Kwon, Ph. D, Study Director — GL PharmTech Corp.
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea